CLINICAL TRIAL: NCT01810250
Title: EVAR Treatment With the Endurant Stent Graft of Challenging Anatomy in Experienced Hands, the Real World Experience
Brief Title: Endurant for Challenging Anatomy: Global Experience Registry
Acronym: EAGLE
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Joep Teijink, MD, PhD, Catharina Ziekenhuis Eindhoven
Other Study IDs: EAGLE Registry
Record Dates: First submitted 2013-02-12; First posted 2013-03-13 (Estimated); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Abdominal Aortic Aneurysms With Challenging Anatomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Abdominal Aortic Aneurysm (Challenging anatomy): Endovascular aneurysm repair
  Interventions: Device: Endurant Stent Graft

INTERVENTIONS:
Device: Endurant Stent Graft

SUMMARY:
The Department of Vascular Surgery at Catharina Hospital Eindhoven, The Netherlands initiates the Endurant for Challenging Anatomy: Global Experience (EAGLE) Registry. The aim of this study is to collect clinical information on the performance of the Endurant Stent Graft System for endovascular repair in anatomically challenging aneurysms, and to critically assess whether the current guidelines for anatomic eligibility to endovascular treatment with this system are still applicable. This study aims at creating a database that can be pooled/ compared with the ENGAGE database.

This study aims at answering two major questions:

1. Is the technical success rate of successful delivery and deployment of the Endurant (II) similar in anatomically challenging aneurysm?
2. Is the successful treatment rate comparable in anatomically challenging aneurysms, or does treatment of these aneurysms lead to more complications and reinterventions?

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years or minimum age as required by local regulations
* Indication for elective EVAR
* Challenging AAA anatomy
* Intention to electively implant the Endurant or Endurant II Stent Graft System©
* Signed informed consent form

Exclusion Criteria:

* Subjects with intolerance to contrast media
* Chimneys or fenestrated device procedures
* High probability of non-adherence to physician's follow-up requirements
* Current participation in a concurrent trial that may confound study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with abdominal aortic aneurysms (AAAs) with challenging anatomy defined by having one or more of the following measurements:
  * Proximal necks 5 - 10mm in combination with < 60 degrees infrarenal AND < 45 degrees suprarenal angulation
  * Proximal necks 10 - 15mm in combination with 60 degrees - 75 degrees infrarenal AND < 60 degrees suprarenal angulation OR in combination with < 75 degrees infrarenal AND 45 degrees - 60 degrees suprarenal angulation
  * Proximal necks > 15mm in combination with 75 degrees - 90 degrees infrarenal AND < 75 degrees suprarenal angulation OR in combination with < 90 degrees infrarenal AND 60 degrees - 75 degrees suprarenal angulation
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-11; Primary Completion 2018-01 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Clinical success | 12 months
  Freedom from:
  * Increase of AAA diameter > 5 mm (1 month measurement as baseline)
  * Type I&III endoleaks
  * Aneurysm rupture
  * Conversion to surgery
  * Stent graft migration (>10mm) resulting in SAE or reintervention
  * Stent graft occlusion

SECONDARY OUTCOMES:
Helath Related Quality of Life Scores | 12 months
  EQ-5D VAS EQ-5D index

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Ziekenhuis, Eindhoven, North Brabant, Netherlands